CLINICAL TRIAL: NCT05285631
Title: Early Prediction of ICD Candidacy After Anterior Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Taha Salah, Principal Investigator, Aswan University
Other Study IDs: EPIC-Anterior-MI
Record Dates: First submitted 2022-02-11; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Anterior MI
MeSH Terms: conditions — Anterior Wall Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Speckle tracking echocardiography (STE) — Two-dimensional (2D) and 3D STE are based on the quantitative analysis of spatial dislocation (tracking) of acoustic markers (""speckles"") generated by the interaction between the ultrasound beam and myocardial fibers during the cardiac cycle.

SUMMARY:
Despite the advances of pharmacologic and interventional therapies, sudden (or arrhythmic) cardiac death remains very high in the early weeks-to-months after an acute myocardial infarction (MI).The majority of cardiac arrests occur in patients who have large infarctions resulting in extensive myocardial damage, which is translated into lower left ventricular ejection fraction (LVEF). Hence, low LVEF remains -to the current time- the most robust predictor for post MI sudden (and presumably arrhythmic) death; and is the determinant for implantable cardioverter defibrillator (ICD) candidacy for primary prevention as per clinical practice guidelines.ICD significantly and effectively reduced ventricular arrhythmia (VA)-mediated cardiac deaths among these patients.

DETAILED DESCRIPTION:
Although the majority of deaths after acute MI occurs in the earlier weeks, however, causes of deaths were almost split between arrhythmic and non-arrhythmic deaths. In the large study conducted by Solomon et al., sudden cardiac death (SCD) was responsible for around 40% of the total mortality.Similarly, arrhythmic death counted for 52% and 49% of the total mortality encountered in the randomized control trial testing role of wearable cardioverter vest in the therapy and control groups respectively, where the remainder were non-arrhythmic (and thus considered non-preventable) deaths.Probably, this fact remains the main driver for the guidelines" writers to label implanting an ICD for primary prevention during the first 90 days after revascularization for MI as class III [contraindicated - no benefit].The large number of potentially preventable SCD triggered investigators to challenge the guidelines" recommendations. At least 3 large, randomized control trials (RCT) tested ICD implantation early prior establishing guidelines-recommended time range; 40 days after MI and/or 90 days after optimal therapy including revascularization.

In the DINAMIT RCT, recruiting 332 patients in the ICD arm vs. 342 in the control arm, ICD significantly reduced arrhythmic death (hazard ratio (HR) 0.42, 95% confidence interval (CI) 0.22 to 0.83;P=0.009). Yet, unfortunately, this benefit was mitigated by the increased non arrhythmic death in the ICD group.Likewise, in the IRIS multicenter RCT, 898 acute MI patients were recruited (445 in the ICD vs 453 in the control arm), ICD significantly reduced SCDs ((27 vs. 60; HR, 0.55; 95% CI, 0.31 to 1.00; P = 0.049)), however, overall mortality was similar between the 2 groups.The third and most recent RCT, "Defibrillator After Primary Angioplasty", the DAPA trial, was published late in 2020.10 Probably reflecting the recent advances in pharmacologic therapies for heart failure and reduced ejection fraction (HFrEF) in the past years, the DAPA trial at its early and long-term follow up reports found that ICD significantly reduced both arrhythmic and all-cause deaths when implanted early to selected patients after primary angioplasty.This unsettled argument between accelerated vs. delayed implantation of ICD for potential candidates after MI sparked for the VEST investigators to randomly assign post MI patients to either Wearable Cardioverter Defibrillator (WCD) plus medical therapy vs. medical therapy alone to test if the wearable device can effectively prevent SCDs during this high risk period.7 Nevertheless, compliance to the WCD was very poor. Despite instructions to wear the device for more than 90% of the time, 43 patients (around 3%) never wore the device and mean ± standard deviation of device wearing time was 14.0±9.3 hours per day, with decreasing use over time. Thus, 75% of the deaths in the device arm occurred while not wearing the vest with strong concerns that the majority of these could have been prevented.Overall, WCD could not effectively reduce death in patients with LVEF ≤ 35% early after MI in this study.Echocardiography has a critical impact on diagnostic and therapeutic decisions in the settings of acute MI. According to the current guidelines, echocardiography-derived LVEF after 90 days of revascularization remains the single most accepted determinant for ICD candidacy. However, there are many limitations in early predicting the LVEF value at the defined time.In the large study conducted by Brooks et al., recruiting patients reduced <35% LVEF acutely post MI with; it was shown at 90 days that only 43% had unchanged LVEF (<35%), while 31% and 26% of the patients have their EF recovered to 36-49% and > 50% respectively. This clearly demonstrates that more than half of the patients with baseline LVEF < 35% had improved at 90 days after revascularization to above the cut-off for ICD eligibility.Speckle tracking echocardiography (STE) have shown great value in improving accuracy of standard echocardiographic assessments.

Two-dimensional (2D) and 3D STE are based on the quantitative analysis of spatial dislocation (tracking) of acoustic markers (""speckles"") generated by the interaction between the ultrasound beam and myocardial fibers during the cardiac cycle.18-20 Global longitudinal strain (GLS) assessed by STE has shown an incremental value beyond traditional echo parameters for risk stratification after AMI.The value of STE to early elicit myocardial structural and functional abnormalities have been shown in many conditions to be more sensitive that the traditional LVEF. This fact elected STE as an accepted sensitive marker to detect myocardial abnormalities before LVEF starts to deviate from normal values such as screening for chemotherapy induced cardiomyopathy.22 An additive role for STE to early identify patients with irreversible myocardial damage contrasted to those with transient/reversible systolic dysfunction can help in earlier patients stratification to receive timed appropriate therapies.Therefore, development of a stratification tool involving advanced imaging modalities besides clinical and laboratory variables that can be utilized to early identify patients eligible for ICD primary prevention therapy can be extremely beneficial to avoid many preventable cardiac deaths in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years. Both genders are eligible.

  * Patients with diagnosis of an acute anterior STEMI and revascularized with successful primary percutaneous coronary intervention (PCI) within 24 hours.
  * LVEF < 40 % assessed by Bi-plane Simpsons rule within 48 hour post PCI.

Exclusion Criteria:

* ● Refusal to participate in the study.

  * Patients with existing ICD or pacemakers.
  * Qualifying ICD for secondary prevention.
  * Known to have LVEF ≤ 40% prior to the index MI.
  * Previous PCI to Left anterior Descending artery (LAD).
  * Previous or being scheduled for CABG within ≤ 3 months.
  * Known to have limited life expectancy (less than 1-year) prior to the index MI.
  * Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting by acute anterior myocardial infarction, with baseline echocardiographic assessment demonstrating LVEF < 40%.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Early prediction of ICD candidacy in anterior STEMI patients by speckle tracking echocardiography | 90 days
  Early prediction of ICD candidacy (EF < 35% after 90 days) by speckle tracking echo performed at baseline and at 30 days

SECONDARY OUTCOMES:
ICD candidacy prediction scores | 90 days
  Development of prediction models for ICD candidacy that can be applied shortly after anterior MI integrating speckle tracking echo, demographic features and comorbidity indices.